CLINICAL TRIAL: NCT03926468
Title: Genetic Profiling by Liquid Biopsy for Initial Characterization and Response Monitoring of Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Liquid Biopsy in Head and Neck Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T17/2019
Record Dates: First submitted 2019-03-14; First posted 2019-04-24 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Liquid biopsy; FDG PET-CT
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating tumor DNA (ctDNA) collected from venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — Before onset of treatment, cell-free DNA (cfDNA) is extracted from venous blood sample for next-generation DNA sequencing (NGS) using a commercially available platform (Roche Foundation ACT) For this purpose, 4 x 10 ml of venous blood will be collected from each patient. Two tubes (Streck) will be sent to service provider (Roche), one tube will be used for droplet digital polymerase chain reaction (ddPCR, QX200 Droplet Digital PCR System, BioRad) and ddPRC/NGS analyses and one is collected and stored in Auria Biobank (www.auria.fi) for possible future analyses.

SUMMARY:
Overall survival of patients with head and neck squamous cell carcinoma (HNSCC) remains unsatisfactory due to often advanced clinical stage at diagnosis and high rate of recurrence and second primaries. About 75 % of patients with localized HNSCC are expected to show circulating tumor DNA (ctDNA) pre-treatment. ctDNA reflects tumor genome and disease burden and is termed 'liquid biopsy' (LB) when collected through venous bloodstream. LB has potential to assist in early diagnosis of recurrence and progression, and prediction of response to targeted therapeutic agents. Increased metabolic activity measured in positron emission tomography-computed tomography (PET-CT) is currently the most sensitive technique to detect residual cancer or progression of HNSCC after curative treatment. High metabolically active tumor volume (MTV) is associated with treatment resistance and shows independent prognostic significance. The objective is (i) to investigate whether MTV detected with PET-CT correlates to the pattern and amount of genetic alterations in ctDNA of patients with HNSCC referred to radio- (chemo)therapy (RT/CRT). Another objective is (ii) to determine sensitivity of LB compared to PET/CT in detecting residual tumor 3 months after completion of RT/CRT. Third (iii), genetic landscape in LB and fresh tumor samples will be evaluated to detect resistance genes and targets for immunotherapy and surveillance post-treatment. This prospective study includes 30 patients with stage III/IV HNSCC. Before onset and 3 months from RT/CRT, LB is obtained for next-generation DNA sequencing using a commercial platform. ctDNA and digital droplet PCR will be quantified and compared to MTV in simultaneously acquired PET-CT. The investigators hypothesize that LB could assist or replace PET/CT in response monitoring and detection of recurrence after RT/CRT.

DETAILED DESCRIPTION:
Background

Head and neck squamous cell carcinoma (HNSCC) stands as the sixth most common cancer worldwide. The overall 5-year survival is approximately 50 % due to often advanced clinical stage at diagnosis, high rate of treatment resistance, and high incidence of second cancers. Currently there are no useful biomarkers for surveillance or diagnosis of recurrent HNSCC.

Liquid biopsy (LB)

Circulating tumor DNA (ctDNA) is tumor-derived fragmented DNA circulating freely in the bloodstream. Apoptosis and necrosis due to rapid cell growth and increased cell turnover contribute to release of ctDNA in circulation of patients with cancer even without disseminated disease. ctDNA reflects tumor genome and may also reflect disease burden. Due to these properties and easy accessibility collection of ctDNA through venous blood has been termed as 'liquid biopsy'. Approximately 75-90 % of patients with localized or untreated HNSCC are expected to show ctDNA pre-treatment.

Applications of liquid biopsy in HNSCC

Potential clinical applications of liquid biopsy (LB) are manifold and include diagnosis of recurrence or progression, and disease surveillance. While ctDNA contains the same mutations present in original tumor, LB can be used to guide targeted therapies if local treatment is not feasible. In HNSCC, these features render study of LB attractive since early diagnosis of treatment failure increases possibilities for curative approach. ctDNA reflects tumor heterogeneity and findings in surveillance samples are more likely to characterize resistant subpopulations compared to pre-treatment changes. Recently, immune checkpoint inhibition with monoclonal antibodies against programmed cell death (PD-1) have demonstrated activity against recurrent or metastatic HNSCC. LB together with evaluation of expression of PD-1 ligand (PD-L1) can assess mutational load thus assisting in screening patients who may benefit from immunotherapy.

Metabolic imaging - current standard for detection of recurrent HNSCC

Increased metabolic activity detected in positron emission tomography-computed tomography (PET-CT) is currently the most sensitive technique to detect residual cancer or progression of HNSCC after curative treatment. High metabolically active tumor volume (MTV) is associated with treatment resistance and shows independent prognostic significance. While PET-CT shows excellent sensitivity, it may lead to false positive findings caused by inflammation or other conditions having increased cellular metabolic rate. Furthermore, metabolic imaging does not elucidate resistance mechanisms nor does it assist in planning of targeted treatments. Whether LB could assist or replace PET/CT in response monitoring and detection of recurrence remains thus far unknown.

Study objectives

i) To investigate whether MTV detected in PET-CT correlates to pattern and amount of genetic alterations in ctDNA of patients with HNSCC referred to radiotherapy (RT) or chemoradiotherapy (CRT) ii) To determine whether LB is more sensitive than PET/CT in detecting residual tumor three months after completion of RT or CRT iii) To evaluate exhaustive genetic landscape of patients with locally advanced HNSCC in order to characterize resistance or target genes for alternative treatments including (but not limited to) immunotherapy, antibodies against epidermal growth factor receptor (EGFR), and hypoxia- and virus-activated compounds iv) To validate a novel digital droplet polymerase chain reaction (PCR) technique for non-invasive surveillance of patients at high risk for recurrence of HNSCC

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed head and neck squamous cell carcinoma (HNSCC)
* WHO performance status 0-2
* clinical stage III patients with bulky T3 primary +/- neck metastasis
* all stage IV patients
* referral to definitive radiotherapy or chemoradiotherapy or multimodality treatment

Exclusion Criteria:

* patients who are not able to sign written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed HNSCC referred to curative multimodality treatment in Hospital District of Southwest Finland
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of circulating tumor DNA (ctDNA) in venous blood sample: Baseline | Baseline
  Measurement of ctDNA with a novel droplet digital polymerase chain reaction (ddPCR)
Diagnostic performance of circulating tumor DNA (ctDNA) in venous blood sample: 3-month follow-up | 3-months after completion of therapy (approximately 6 months post-baseline)
  Measurement of ctDNA with a novel droplet digital polymerase chain reaction

CONTACTS AND LOCATIONS:
Overall Officials: Heikki RI Minn, Prof., MD, Principal Investigator — Head, Department of Oncology and Radiotherapy
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Mehanna H, Wong WL, McConkey CC, Rahman JK, Robinson M, Hartley AG, Nutting C, Powell N, Al-Booz H, Robinson M, Junor E, Rizwanullah M, von Zeidler SV, Wieshmann H, Hulme C, Smith AF, Hall P, Dunn J; PET-NECK Trial Management Group. PET-CT Surveillance versus Neck Dissection in Advanced Head and Neck Cancer. N Engl J Med. 2016 Apr 14;374(15):1444-54. doi: 10.1056/NEJMoa1514493. Epub 2016 Mar 23. PMID 27007578
- [Background] Castelli J, De Bari B, Depeursinge A, Simon A, Devillers A, Roman Jimenez G, Prior J, Ozsahin M, de Crevoisier R, Bourhis J. Overview of the predictive value of quantitative 18 FDG PET in head and neck cancer treated with chemoradiotherapy. Crit Rev Oncol Hematol. 2016 Dec;108:40-51. doi: 10.1016/j.critrevonc.2016.10.009. Epub 2016 Oct 29. PMID 27931839